CLINICAL TRIAL: NCT01707303
Title: Effect Of Acute Inflammatory Mediators On Duration Of Functional Limitations In Patients With Acute Respiratory Failure, A Randomized, Controlled Pilot Study of Early ICU Rehabilitation Strategies
Brief Title: Effect Of Acute Inflammatory Mediators On Functional Limitations In Patients With Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00000240
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Acute Respiratory Failure
Keywords: ICU; Critical Care; Intensive Care; Critical Illness; Acute Respiratory Failure; Mechanical Ventilation; Physical Therapy; Strength; Functional Status; Short Physical Performance Battery
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other): Usual hospital rehabilitative services
  Interventions: Other: Usual Care
- Early ICU Rehabilitation Strategy (Experimental): Early ICU physical therapy will be applied in this arm
  Interventions: Other: Early ICU rehabilitation strategies

INTERVENTIONS:
Other: Early ICU rehabilitation strategies — Physical therapy - standard; Physical therapy, progressive resistance training for 2nd physical therapy session in Cohort II
  Other Names: Cohort I will receive one physical therapy session per day; Cohort II will receive 2 physical therapy sessions per day.
  Arms: Early ICU Rehabilitation Strategy
Other: Usual Care — All typically applied hospital rehabilitative services applied in the usual fashion
  Other Names: Usual Hospital Rehabilitative Services
  Arms: Usual Care

SUMMARY:
This is a randomized, controlled, pilot study of two separate Cohorts of patients from the intensive care unit. Cohort I will enroll 50 patients and randomize to receive one physical therapy session per day or receive usual ICU care. Cohort II, will enroll an additional 50 patients and randomize to receive either two physical therapy sessions per day or usual care. Outcome will be length of hospital stay measured in days. Secondary outcomes will be mortality, ventilator days, ICU days, and for Cohort II, grip strength, dynamometer strength assessments and the short physical performance battery (SPPB). Study subjects will have blood for cytokine analysis through their first week of study.

ELIGIBILITY:
Inclusion Criteria:

• Mechanically ventilated via an endotracheal tube or mask

Exclusion Criteria:

* Inability to walk without assistance prior to acute ICU illness (use of a cane or walkers not exclusions)
* Cognitive impairment prior to acute ICU illness (non-verbal)
* Preadmit immunocompromised (>prednisone 20 mg/d for 2 wks)
* Acute stroke
* Body mass index (BMI) >45
* Neuromuscular disease that could impair weaning (myasthenia gravis, ALS, Guillain-Barre)
* Hip fracture, unstable cervical spine or pathological fracture
* Mech vent >48 hours prior to transfer from an outside facility
* Current hospitalization or transferring hospital stay >72 hours
* CPR on admission, DNR on admission
* Hospitalization within 30 days prior to admission
* Cancer therapy within last 6 months
* Re-admission to ICU within current hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay, days | The participants will be followed for the duration of the hospitalization, an expected average of 3 weeks.
  Hospital stay measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Peter E. Morris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No